CLINICAL TRIAL: NCT03377231
Title: Assessment of Efficacy, Safety and Tolerability of Stratamark® (Innovative Self-drying Silicone Gel) in the Treatment and Prevention of Striae Distensae
Brief Title: Prevention and Treatment of Stretch Marks With Stratamark™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stratpharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SPASK01AU001; SSA/13/WCHN/42 (Other: WCHN Human Research Ethics Committee)
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Stretch Mark
Keywords: Pregnancy, Striae gravidarum, Striae distensae, Women's health
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Intervention Model Description: The study involved the use of Stratamark® in prevention and treatment of stretch marks in 2 study arms.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevention (Experimental)
  Interventions: Device: Stratamark®
- Treatment (Experimental)
  Interventions: Device: Stratamark®

INTERVENTIONS:
Device: Stratamark® — Film-forming dressing for the prevention and treatment of stretch marks.

SUMMARY:
Stretch marks (striae distensae) are a form of scarring that is a natural result of pregnancy, obesity and in some instances occur due to puberty or steroid use. For some people, the stretch marks do not cause a problem, but in many circumstances they can cause physical symptoms such as itchiness, tenderness and pain. For many people stretch marks are also embarrassing and can have detrimental effects on a patient's mood and self-esteem. Stretch marks that result from pregnancy most commonly occur on the abdomen, breasts and thighs.

Topical silicone gel was developed nearly thirty years ago to be used in the treatment of widespread hypertrophic scars (abnormal scars, which may be red or raised/depressed itchy or painful). Since this time it has been used successfully on most scar types. . Since stretch marks are a form of scarring it is thought that topical silicone gel may be helpful for this scar type also. Stratamark™ has been developed using different forms of silicone polymers, in a gel format, that dries to form a very thin and flexible silicone gel sheet making it a convenient therapy for the treatment and prevention of stretch marks.

The aim of this clinical research study is to prove or disprove the efficacy, safety and tolerability of Stratamark™ in the prevention and treatment of stretch marks. In addition, the knowledge gained from this study may be of benefit to many future patients

ELIGIBILITY:
Prevention arm - Inclusion Criteria:

* Healthy pregnant woman (nulliparous or multiparous) entering into their third trimester (26-28 weeks, visit 1)
* Not having striae on their abdomen at the time of trial enrollment

Prevention arm - Exclusion Criteria:

* Any significant medical or surgical conditions
* Current medications liable to interfere with study results or change the skin's response to therapy

Treatment arm - Inclusion Critera:

• Confirmed SD on their abdomen post-delivery

Treatment arm - Exclusion Criteria:

* Any significant medical or surgical conditions
* Current medications liable to interfere with study results or change the skin's response to therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 272 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2016-05-16 (Actual); Study Completion 2016-05-16 (Actual)

PRIMARY OUTCOMES:
Product efficacy in prevention of stretch marks | 5 months
  Investigator-assessed prevalence of stretch marks in the patients treated with Stratamark vs. a literature-based control group.
  Measurement tool: dichotomous scale for the occurrence of stretch marks (0 no stretch marks - 1 appearance of stretch marks).
Product efficacy in treatment of stretch marks | 6 months
  Investigator-assessed improvement in stretch marks severity of patients treated with Stratamark from baseline to last assessment.
  Measurement tool: likert scale for stretch marks severity (0 to 6 - 0 being no stretch marks and 6 being severe).

SECONDARY OUTCOMES:
Severity of stretch marks developed in prevention | 5 months
  Investigator-assessed severity of stretch marks developed in prevention patients.
  Measurement tool: likert scale for stretch marks severity (0 to 6 - 0 being no stretch marks and 6 being severe).
Patient product evaluation in prevention of stretch marks | 5 months
  Patient-perceived product efficacy, tolerability, ease of use and feel on skin at trial completion.
  Measurement tool: likert scale for product evaluation (0 to 4 - 0 being unsatisfactory and 4 being excellent).
Product efficacy in treatment of stretch marks | 6 months
  Investigator-assessed improvement in stretch marks color of patients treated with Stratamark from baseline to last assessment.
  Measurement tool: likert scale for stretch marks color assessment (-4 to +4 - -4 being stark white compared to surrounding skin and +4 being purple).
  0 being normal skin color, is considered to be the optimal value.
Product efficacy in treatment of stretch marks | 6 months
  Investigator-assessed improvement in stretch marks pruritus of patients treated with Stratamark from baseline to last assessment.
  Measurement tool: likert scale for stretch marks pruritus assessment (0-10 - 0 being no pruritus and 10 being worst possible pruritus).
Patient product evaluation in treatment of stretch marks | 6 months
  Patient-perceived product efficacy, tolerability, ease of use and feeling on skin at trial completion.
  Measurement tool: likert scale for product evaluation (0 to 4 - 0 being unsatisfactory and 4 being excellent).
Patient evaluation of stretch marks in treatment | 6 months
  Patient-perceived change in color and noticeability of stretch marks at trial completion.
  Measurement tool: likert scale for stretch marks patient evaluation (-4 to +4 - -4 being much worse and +4 being cleared).